CLINICAL TRIAL: NCT06707220
Title: The Türkiye Heart Failure (TURK-HF) Registry
Brief Title: The Türkiye Heart Failure Registry
Acronym: TURK-HF
Status: Recruiting | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Umut Kocabas, Medical Doctor, Baskent University
Other Study IDs: KA23/429
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Heart failure medication — Treated with optimal guideline-directed medical therapy

SUMMARY:
A comprehensive understanding of the socio-demographic, clinical, and biological characteristics of patients with heart failure is essential to develop novel strategies for improving outcomes. The identification of the barriers to guideline-directed medical therapy implementation in a real-world setting is critical to decreasing the risk of heart failure hospitalization and mortality. A comprehensive and well-designed heart failure registry can determine the clinical characteristics of patients with heart failure, identify patient, physician, and healthcare system-related factors for the non-use of evidence-based therapies, and improve the implementation of guideline-directed medical therapy. It should be noted that the number of heart failure registries that enroll patients with de novo heart failure, chronic heart failure (outpatients), and worsening of heart failure (hospitalized or treated in the emergency department), with all three relevant ejection fraction categories (heart failure with reduced ejection fraction, heart failure with mildly-reduced ejection fraction, and heart failure with preserved ejection fraction), is limited. Furthermore, only a few registries assess detailed aspects of guideline adherence, treatment decisions, and both in-hospital and long-term outcomes. Therefore, the Türkiye Heart Failure (TURK-HF) registry has been designed to address this gap in knowledge about the identification, management, and long-term prognosis of patients with heart failure in a real-world setting.

ELIGIBILITY:
Inclusion Criteria: Presence of heart failure -

Exclusion Criteria: Age <18 years

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The only inclusion criterion for the Türkiye Heart Failure (TURK-HF) registry is the presence of heart failure, as determined by an investigator, and the only exclusion criterion is age <18 years. All patients will be eligible for enrollment regardless of their ejection fraction and whether they have pre-existing chronic or de novo heart failure. All patients will be enrolled in the study, regardless of their clinical status. This encompasses both those presenting for a non-urgent outpatient visit with stable signs and symptoms and those requiring urgent care with worsening of heart failure. Worsening heart failure is defined as worsening symptoms and signs of heart failure in patients with pre-existing heart failure, requiring hospitalization and/or intravenous diuretic therapy. All study participants must provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Heart failure hospitalization | From enrollment to the end of follow-up period at 12 months
Cardiovascular mortality | From enrollment to the end of follow-up period at 12 months
Composite of heart failure hospitalization and cardiovascular mortality | From enrollment to the end of follow-up period at 12 months

SECONDARY OUTCOMES:
All-cause mortality | From enrollment to the end of follow-up period at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kocabas U, Ergin I, Yavuz V, Altin C, Kaplan M, Yilmaz Oztekin GM, Dogdus M, Murat S, Murat B, Kivrak T, Karabulut D, Kaya E, Ozdemir IH, Yildiz C, Salkin FO, Ozcalik E, Polatkan SG, Cakan F, Sen T, Karabulut U, Cakal S, Oflar E, Sinan UY, Yenercag M, Turk UO. Real-world data on Empagliflozin and Dapagliflozin use in patients with HEART failure: The RED-HEART study. ESC Heart Fail. 2025 Feb;12(1):434-446. doi: 10.1002/ehf2.15049. Epub 2024 Sep 28. PMID 39340234
- [Background] Kocabas U, Ergin I, Kivrak T, Yilmaz Oztekin GM, Tanik VO, Ozdemir I, Avci Demir F, Dogdus M, Sen T, Altinsoy M, Ustundag S, Urgun OD, Sinan UY, Uygur B, Yeni M, Ozcalik E. Prognostic significance of medical therapy in patients with heart failure with reduced ejection fraction. ESC Heart Fail. 2023 Dec;10(6):3677-3689. doi: 10.1002/ehf2.14559. Epub 2023 Oct 7. PMID 37804042
- [Background] Kocabas U, Kivrak T, Yilmaz Oztekin GM, Tanik VO, Ozdemir IH, Kaya E, Yuce EI, Avci Demir F, Dogdus M, Altinsoy M, Ustundag S, Ozyurtlu F, Karagoz U, Karakus A, Urgun OD, Sinan UY, Mutlu I, Sen T, Astarcioglu MA, Kinik M, Tok OO, Uygur B, Yeni M, Alan B, Dalgic O, Sariturk C, Altay H, Pehlivanoglu S. Adherence to guideline-directed medical and device Therapy in outpAtients with heart failure with reduced ejection fraction: The ATA study. Anatol J Cardiol. 2020 Jul;24(1):32-40. doi: 10.14744/AnatolJCardiol.2020.91771. PMID 32628147